CLINICAL TRIAL: NCT05716750
Title: Serum Prolidase Activity and the Role of Leptin in Osteomalacia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TUĞBA ŞAHBAZ (Other)
Responsible Party: Sponsor-Investigator, TUĞBA ŞAHBAZ, assist. prof. dr, University of Beykent
Organization: University of Beykent (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAEK/2022.12.233
Record Dates: First submitted 2023-01-09; First posted 2023-02-08 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Osteomalacia
MeSH Terms: conditions — Osteomalacia | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Osteomalasia (Other): Our study, which is the only group planned prospectively, aims to compare clinical and laboratory data and serum prolidase activity and leptin levels in 38 patients diagnosed with osteomalacia after and before 8 weeks of 50,000 IU D vit treatment.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — 50,000 IU vit D treatment for 8 weeks
  Other Names: vit D treatment

SUMMARY:
Evaluation of the change of serum Prolidase and Leptin values in the diagnosis and follow-up of osteomalacia and its clinical usability

DETAILED DESCRIPTION:
Osteomalacia describes a bone disorder in adults that is usually caused by long-term vitamin D deficiency. Osteomalacia, a metabolic bone disease characterized by impaired mineralization of the bone matrix.Not a single laboratory finding is specific to osteomalacia.The relationship between collagen and prolidase activity has been observed during fibrotic processes, where an increase in prolidase activity is accompanied by an increase in tissue collagen deposition. It has also been suggested that serum activity is increased in metabolic bone diseases.Leptin is a 16 kDa peptide hormone. It is a member of the long chain helical cytokine family, which is mainly produced by fat cells and proportional to the size of the stored fat. Leptin affects bone remodeling by reducing the activity of osteoclasts and thus participates in the pathogenesis of osteoporosis. In the light of these studies, the investigators planned our study according to the clinical significance of serum prolidase activity in osteomalacia and the place of leptin in osteomalacia.

ELIGIBILITY:
Inclusion Criteria:

* Among the patients who applied to the outpatient clinic, those with clinical complaints of osteomalacia (diffuse pain, fatigue, rapid fatigue, proximal extremity weakness, etc.)
* 25 0H vit. D level of 10ng/ml and below

Exclusion Criteria:

* Other metabolic and endocrine bone diseases (secondary osteoporosis, paget hast, osteogenesis imperfecta, osteomyelitis etc.)
* Patients who have previously received treatment for low vitamin d
* Those with low vitamin D levels due to liver or kidney failure
* Those who receive treatment for tumor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum Prolidase activity | 8 weeks
  Prolidase activity
Serum Leptin | 8 weeks
  Leptin

IPD SHARING:
Plan to Share IPD: No